CLINICAL TRIAL: NCT06089993
Title: Impact of Acute Resistance Exercise on Taste Perception and Appetite Response to Plant Protein in Resistance Trained Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Katy Horner, Lecturer in Sport and Exercise Science, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: LS-22-30-Horner
Record Dates: First submitted 2023-03-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Appetite; Taste, Altered; Exercise
Keywords: protein; plant protein; soy protein; hemp protein; brown rice protein; pea protein; whey protein; taste perception; taste; appetite; sensory perception; Visual Analogue Scale; Likert Scale; strength training; resistance training
MeSH Terms: conditions — Dysgeusia; Motor Activity | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Resistance exercise involves 4 exercises (bench pull, bench press, leg extension and unilateral leg press), that are performed at 75% of maximum, determined from 3-RM test.
  Interventions: Other: Exercise
- Rest (Experimental): One hour rest.
  Interventions: Other: Rest

INTERVENTIONS:
Other: Exercise — The total volume of exercise is 40 repetitions of each of the 4 exercises. The participant is instructed to perform a maximum of 10 repetitions each set, with 1'30'' rest between sets and between exercises. The researcher provides instructions and verbal encouragement. The total duration of the exercise bout is between 1 hour and 1 hour and 15 minutes.
  Part 1: Before and after the exercise condition the participant is sampling 8 different samples: (1) sucrose (2) umami (3) soy protein (4) pea protein (5) hemp protein (6) brown rice (7) whey protein and (8) apple juice.
  All protein sources are 3 grams dissolved in 20ml apple juice. Sucrose is 1.66g in 20ml water and umami tastant is 0.09g in 20ml water.
  Part 2: a 30g soy protein bolus in 200ml apple juice is given to the participant. After 1 hour energy intake is assessed with an ad libitum lunch meal.
  Arms: Exercise
Other: Rest — The participant remains in sedentary activities such as reading or using a laptop.
  Part 1: Before and after the rest condition the participant is sampling 8 different samples: (1) sucrose (2) umami (3) soy protein (4) pea protein (5) hemp protein (6) brown rice (7) whey protein and (8) apple juice.
  All protein sources are 3 grams dissolved in 20ml apple juice. Sucrose is 1.66g in 20ml water and umami tastant is 0.09g in 20ml water.
  Part 2: a 30g soy protein bolus in 200ml apple juice is given to the participant. After 1 hour energy intake is assessed with an ad libitum lunch meal.
  Arms: Rest

SUMMARY:
Some evidence suggests that taste perception might be modulated by physical exercise, with differences observed after aerobic exercise (DOI:10.1093/chemse/23.4.417) and with habitual exercise (DOI:10.3390/nu11010155). However, the effects of resistance exercise on taste perception has not been studied. This knowledge is important as it may impact the acceptability of foods consumed after exercise.

While plant-protein supplement powders are gaining increased popularity, their palatability and, thereby, acceptability may be a shortcoming. This randomised crossover trial aims to investigate (1) the taste perception and acceptability of plant protein supplement powders and (2) whether resistance exercise modulates taste perception and appetite responses to plant protein.

DETAILED DESCRIPTION:
Phase 1 (part 1): A randomised crossover trial, involving 15-20 adult men (aged 18-40 years old). Two conditions (resistance exercise or rest) will be undertaken in randomised order.

Participants will be required to attend three tests visits. The first visit will last approximately 2 hours and involves signing informed consent, body composition assessment (BodPod), strength tests (3-Repetition Maximum) and completion of questionnaires.

The second and third visits are the experimental test visits (exercise or rest) and will last approximately 4 hours each. Individuals will arrive at the laboratory two hours after consuming a standardized breakfast.

Participants will be provided with eight food-grade samples and asked to complete a battery of questionnaires to evaluate taste perception and liking (visual analogue scales (VAS), generalised labelled magnitude scale (gLMS), 9-point Likert scale). The eight samples are: (1) sucrose (2) umami (3) soy protein (4) pea protein (5) hemp protein (6) brown rice (7) whey protein and (8) apple juice. Each sample will be served as a 20-mL-solution. Except for sucrose and umami (in water), the protein-based samples will be served in low sugar apple juice. Subjects will taste the samples in a "sip-and-spit" manner. Each solution will be designated by a 3-digit number and they will be provided in a randomized order.

Participants will then undergo approximately 1 hour of rest (control) or resistance exercise conditions, after which they will repeat an identical tasting session of the 8 samples.

The resistance exercise will be composed of the 4 exercises, that will be performed at a high-to-medium intensity (75% of the maximum calculated), intensity represented by 10 estimated repetitions. Four sets of each exercise will be assisted by the investigator.

Phase 1 (part 2): The second part of each test visit (exercise or rest) involves the participant consuming a soy protein drink (30g soy protein powder, according to most of the manufacturer's recommendation) solubilized in 200ml low-sugar apple juice (to increase palatability). After an hour of rest, the participant will then be served an ad libitum lunch meal (pasta bake with tomato sauce and cheese, strawberry yogurt and water). Appetite will be assessed both during rest and after the lunch meal via VAS.

Saliva samples will also be collected at three time-points during the test visit to provide insight into potential mechanisms contributing to alterations in taste perception and appetite.

Phase 2: Part 1 is extended to 15-20 adult female participants (18-40 years old) to provide insight into any potential sex differences in findings. The eight samples tested are identical except brown rice protein is replaced with clear protein isolate (a form of hydrolysed pea protein).

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: Adult males; Phase 2: Adult females
* Aged between 18 and 40 y.o.)
* Physically active in accordance with IPAQ
* Lifting weights, at least, once a week
* Healthy
* Non-smokers
* BMI between 18 and 30

Exclusion Criteria:

* Phase 1: Females; Phase 2: Males
* Subjects younger than 18 or older than 40 y.o.
* BMI lower than 18 and higher than 30
* Insufficiently active individuals
* Physical active individuals that do not perform a regular strength training
* Having any condition health-related that could preclude both their participation in physical testing and a bout of resistance training
* Taking medications known to impact taste and/or appetite
* Medical condition known to impact taste and/or appetite
* Medical condition linked to cognitive impairment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Part 1: Change in Taste Intensity | 2 hours: (1) baseline sampling session, (2) post-intervention sampling session (i.e. after 1 hour resistance training or rest).
  Taste intensity from Generalised Labelled Magnitude Scale (gLMS)
  Validated 200 millimetre scales will be used to assess intensity of the taste of each sample.
  This scale has anchors located at each end of the scale and along the scale (barely detectable, weak, moderate, strong, very strong, strongest imaginable). On the bottom end of the scale, the extreme negative response (0 mm) is represented, while the top end (200 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.
Part 1: Change in Liking of the samples | 2 hours: (1) baseline sampling session, (2) post-intervention sampling session (i.e. after 1 hour resistance training or rest). Change scores will be compared between exercise and rest condition.
  9-point Likert Scale to rate overall liking of each sample, from 0 (dislike extremely) to 9 (like extremely).
Part 2: Change in Appetite - Composite Appetite Score | 3.5 hours: (1) at participant arrival, (2) after exercise or resting condition (3) immediately after the protein bolus (4) 30 minutes after the protein bolus (5) 60 minutes after the protein bolus (6) after the lunch meal
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to assess appetite, at six (6) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Composite Appetite Score derived from aspects such as hunger, fullness, desire to eat and prospective food consumption will be calculated.
Part 2: Energy Intake | Day 2 and Day 3
  Energy intake measurement. Participants will be given a standardised fixed breakfast to be eaten at home 2 hours prior the testing visit. At the end of the testing visit participants will be served with ad libitum lunch meal in the laboratory. Lunch EI (kilocalories) will be measured objectively, by weighing foods before and after consumption and calculating energy intake based on their nutritional data. EI will be compared between exercise and rest conditions

SECONDARY OUTCOMES:
Part 2: changes in cortisol | 3 hours: (1) immediately after participant arrival, (2) after exercise or rest, (3) 1 hour after exercise or rest (i.e. immediately before the lunch meal)
  Saliva sample will be collected by passive drooling three (3) times.
Part 2: changes in testosterone | 3 hours: (1) immediately after participant arrival, (2) after exercise or rest, (3) 1 hour after exercise or rest (i.e. immediately before the lunch meal)
  Saliva sample will be collected by passive drooling three (3) times.
Part 2: Palatability - Pleasantness | Day 2 and Day 3
  100 millimetre Visual Analogue Scales (VAS) will be used immediately after the protein bolus and the lunch meal. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Data will be compared between exercise and rest conditions.
Part 2: Palatability - Filling | Day 2 and Day 3
  100 millimetre Visual Analogue Scales (VAS) will be used immediately after the protein bolus and the lunch meal. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Data will be compared between exercise and rest conditions.
Part 2: Palatability - Satisfaction | Day 2 and Day 3
  100 millimetre Visual Analogue Scales (VAS) will be used immediately after the protein bolus and the lunch meal. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Data will be compared between exercise and rest conditions.
Part 2: Palatability - Taste | Day 2 and Day 3
  100 millimetre Visual Analogue Scales (VAS) will be used immediately after the protein bolus and the lunch meal. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Data will be compared between exercise and rest conditions.
Part 2: Palatability - Sweet | Day 2 and Day 3
  100 millimetre Visual Analogue Scales (VAS) will be used immediately after the protein bolus and the lunch meal. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Data will be compared between exercise and rest conditions.
Part 2: Palatability - Savoury | Day 2 and Day 3
  100 millimetre Visual Analogue Scales (VAS) will be used immediately after the protein bolus and the lunch meal. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the extreme negative response is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Data will be compared between exercise and rest conditions.
Part 2: Changes in Hunger | 3.5 hours: (1) at participant arrival, (2) after exercise or resting condition (3) immediately after the protein bolus (4) 30 minutes after the protein bolus (5) 60 minutes after the protein bolus (6) after lunch. Mixed model ANOVA will be used.
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, at six (6) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Data will be compared between exercise and rest conditions.
Part 2: Changes in Fullness | 3.5 hours: (1) at participant arrival, (2) after exercise or resting condition (3) immediately after the protein bolus (4) 30 minutes after the protein bolus (5) 60 minutes after the protein bolus (6) after lunch. Mixed model ANOVA will be used.
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, at six (6) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Data will be compared between exercise and rest conditions.
Part 2: Changes in Desire to Eat | 3.5 hours: (1) at participant arrival, (2) after exercise or resting condition (3) immediately after the protein bolus (4) 30 minutes after the protein bolus (5) 60 minutes after the protein bolus (6) after lunch. Mixed model ANOVA will be used.
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, at six (6) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Data will be compared between exercise and rest conditions.
Part 2: Changes in Prospective Food Consumption | 3.5 hours: (1) at participant arrival, (2) after exercise or resting condition (3) immediately after the protein bolus (4) 30 minutes after the protein bolus (5) 60 minutes after the protein bolus (6) after lunch. Mixed model ANOVA will be used.
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to estimate changes in appetite, at six (6) set time points throughout the experimental visit. This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Data will be compared between exercise and rest conditions.
Part 1: Changes in Sensory Perception - Visual Appeal | 2 hours: (1) baseline sampling session, (2) post-intervention sampling session (i.e. after 1 hour resistance training or rest)
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to assess sensory perception during two sampling session (8 times each sampling session). This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends. Change scores will be compared between exercise and rest conditions.
Part 1: Changes in Sensory Perception - Smell | 2 hours: (1) baseline sampling session, (2) post-intervention sampling session (i.e. after 1 hour resistance training or rest)
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to assess sensory perception during two sampling session (8 times each sampling session). This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Change scores will be compared between exercise and rest conditions.
Part 1: Changes in Sensory Perception - Taste | 2 hours: (1) baseline sampling session, (2) post-intervention sampling session (i.e. after 1 hour resistance training or rest)
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to assess sensory perception during two sampling session (8 times each sampling session). This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Change scores will be compared between exercise and rest conditions.
Part 1: changes in Sensory Perception - Aftertaste | 2 hours: (1) baseline sampling session, (2) post-intervention sampling session (i.e. after 1 hour resistance training or rest)
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to assess sensory perception during two sampling session (8 times each sampling session). This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Change scores will be compared between exercise and rest conditions.
Part 1: Changes in Sensory Perception - Palatability | 2 hours: (1) baseline sampling session, (2) post-intervention sampling session (i.e. after 1 hour resistance training or rest)
  Validated 100 millimetre Visual Analogue Scales (VAS) will be used to assess sensory perception during two sampling session (8 times each sampling session). This VAS has anchors located at each end of the scale. On the left end of the scale, the extreme negative response (0 mm) is represented, while the right end (100 mm) represents the positive response. Participants mark along the line where it most represents their subjective perception between both ends.Change scores will be compared between exercise and rest conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Ireland